

# **Statistical Analysis Plan**

Version 3.0 01 October 2021

**Protocol Title:** Prospective, Phase 3, multi center, single-arm, imaging study investigating the safety and diagnostic performance of rhPSMA-7.3 (<sup>18</sup>F) PET ligand in men with newly diagnosed prostate cancer

**Protocol Number: BED-PSMA-301** 

Compound Number: Flotufolastat (18F) injection

**Short Title:** LIGHTHOUSE

Sponsor Name: Blue Earth Diagnostics Ltd.

Legal Registered Address: Magdalen Centre, Robert Robinson Avenue, The

Oxford Science Park. Oxford, OX4 4GA, UK

**IND** 141,561

**NCT** 04186819

Blue Earth Diagnostics BED-PSMA-301

Statistical Analysis Plan

### **PAREXEL International**

Blue Earth Diagnostics

BED-PSMA-301

A prospective, Phase 3, multi center, single-arm, imaging study investigating the safety and diagnostic performance of rhPSMA-7.3 (<sup>18</sup>F) PET ligand in men with newly diagnosed prostate cancer

Statistical Analysis Plan

Version: 3.0

**PAREXEL Project Number: 245596** 

TP-GDO-WW-016-07.a CONFIDENTIAL **Project Document Version No.** 3.0 Effective Date: 30 Jan 19 **Project Document Effective Date**: Date of last signature Related to: SOP-GDO-WW-019 

Blue Earth Diagnostics BED-PSMA-301

Approved by:

Statistical Analysis Plan

### **SPONSOR SIGNATURE PAGE**

01-Oct-2021

Albert Chau

Date

Director of Biometrics (interim) Blue Earth Diagnostics Ltd.

TP-GDO-WW-016-07.a CONFIDENTIAL **Project Document Version No.** 3.0 Effective Date: 30 Jan 19 **Project Document Effective Date**: Date of last signature Related to: SOP-GDO-WW-019 

Blue Earth Diagnostics BED-PSMA-301

Statistical Analysis Plan

### PAREXEL SIGNATURE PAGE

Signature(s) below confirm that the Statistical Analysis Plan was developed in accordance with SOP-GDO-WW-019 and that it is approved for release.

This document has been approved and signed electronically by the following:

| | Signatory |
|--------|-----------------------------------------------------------------|
| Author | Kees Duineveld Project Role: Biostatistics Lead/Biostatistician |
| | Dogi Closed by |

Signer Name: Kees Duineveld Signing Reason: I am the author of this documen Signing Time: 01-Oct-2021 | 4:09:08 AM PDT AC6BBDD8D7E04E2E9D735FC7C9119C6C

TP-GDO-WW-016-07.a CONFIDENTIAL **Project Document Version No. 3.0** Effective Date: 30 Jan 19 Project Document Effective Date: Date of last signature Related to: SOP-GDO-WW-019

Blue Earth Diagnostics BED-PSMA-301

Statistical Analysis Plan

| TABLE OF | CONTENTS |
|----------|----------|

| LIST OF | ABBREVIATIONS | 7 |
|---|---|---|
| 1 | INTRODUCTION | 9 |
| 2 | STUDY OBJECTIVES | 10 |
| 2.1 | Primary Objective(s) | 10 |
| 2.2 | Secondary Objective(s) | 10 |
| 2.3 | Exploratory Objective(s) | 11 |
| 3 | INVESTIGATIONAL PLAN | 11 |
| 3.1 | Overall Study Design and Plan | 11 |
| 3.2 | Endpoints | 12 |
| 3.2.1 | Primary Efficacy Endpoint | 12 |
| 3.2.2 | Secondary Efficacy Endpoints | 12 |
| 3.2.3 | Exploratory Efficacy Endpoints | 13 |
| 3.2.4 | Safety Variables | 13 |
| 4 | STATISTICAL METHODS | 13 |
| 4.1 | Data Quality Assurance | 13 |
| 4.2 | General Presentation Considerations | 13 |
| 4.3 | Software | 14 |
| 4.4 | Study Patients | 15 |
| 4.4.1 | Disposition of Patients | 15 |
| 4.4.2 | Protocol Deviations | 15 |
| 4.5 | Analysis Sets | 16 |
| 4.6 | Demographic and Other Baseline Characteristics | 17 |
| 4.6.1 | Demographics | 17 |
| 4.6.2 | Baseline conventional imaging | 17 |
| 4.6.3 | Prostate Cancer History | 17 |
| 4.6.4 | Baseline Risk Category | 18 |
| 4.6.5 | Medical history | 19 |
| 4.7 | Prior and Concomitant Medications and Procedures | 19 |
| 4.8 | Exposure and Treatment Compliance | 19 |
| 4.9 | rhPSMA-7.3 ( <sup>18</sup> F) Image reading | 20 |
| 4.10 | Biopsy/Surgery | 20 |
| 4.11 | TNM staging and Gleason score | 21 |
| 4.12 | Standard of Truth | 21 |
| 4.13 | Hemipelvis Region Categorization and Patient Level Categorization | 22 |
| 4.14 | Efficacy Evaluation | 24 |
| 4.14.1 | Analysis and Data Conventions | 24 |
| 4.14.1.1 | Adjustments for Covariates | 24 |
| 4.14.1.2 | Handling of Dropouts or Missing Data | 24 |
| 4.14.1.3 | Interim Analyses | 25 |
| 4.14.1.4 | Examination of Subgroups | 25 |
| 4.14.1.5 | Clustered binary data estimate of variance | 25 |
| | 4.14.1.5.1 Sensitivity | 25 |
| | 4.14.1.5.2 Additional Confidence interval Sensitivity | 26 |
| | 4.14.1.5.3 Specificity | 26 |

TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019 CONFIDENTIAL Project Document Version No. 3.0

Project Document Effective Date: Date of last signature


| | Diagnostics | |
|---|---|---|
| BED-PSM. | | lan |
| 4.14.2 | Primary Efficacy Variable | 26 |
| 4.14.2.1 | Sensitivity Analysis; patients with FN and FP results | 27 |
| 4.14.3 | Secondary Efficacy Variables | 27 |
| 4.14.3.1 | Percentage of patients in whom rhPSMA-7.3 ( <sup>18</sup> F) imaging detects at least one verification | fied |
| | M1 metastasis, as determined by central BIE. | 27 |
| 4.14.3.2 | Percentage of patients with negative conventional imaging for M1 disease in whom | l |
| | rhPSMA-7.3 (18F) PET detects at least one verified M1 metastasis, as determined by | y |
| | central BIE. | 28 |
| 4.14.3.3 | Patient level PPV of rhPSMA-7.3 ( <sup>18</sup> F) PET BIE for N1 and M1 lesions compared to | to |
| | histopathology or confirmatory imaging (M1 lesions only). | 28 |
| 4.14.3.4 | PPV of rhPSMA-7.3 ( <sup>18</sup> F) PET for detecting pelvic LN metastases compared to | |
| | surgical pathology on a patient level in which a FP patient is defined as having at le | ast |
| | one FP region (right or left pelvis), regardless of any coexisting TP findings. | 29 |
| 4.14.3.5 | NPV of rhPSMA-7.3 ( <sup>18</sup> F) PET for detecting pelvic LN metastases compared to | |
| | surgical pathology on a patient level in which a FN patient is defined as having at le | east |
| | one FN region (right or left pelvis), regardless of any coexisting TN findings. | 29 |
| 4.14.3.6 | Upstaging | 29 |
| 4.14.3.7 | Kappa statistic for the agreement between and within blinded independent readers of | |
| | the interpretation of rhPSMA-7.3 ( <sup>18</sup> F) scans. | 30 |
| | 4.14.3.7.1 Inter-reader agreement analysis | 30 |
| | 4.14.3.7.2 Intra-reader agreement analysis | 30 |
| 4.14.4 | Exploratory Efficacy Variables | 30 |
| 4.14.4.1 | Diagnostic performance (sensitivity and specificity) of rhPSMA-7.3 ( <sup>18</sup> F) PET for | |
| | detecting pelvic LN metastases compared to surgical pathology on a regional level. | 30 |
| 4.15 | Safety Evaluation | 31 |
| 4.15.1 | Adverse Events | 31 |
| 4.15.2 | Deaths, Serious Adverse Events, and Other Significant Adverse Events | 32 |
| 4.15.3 | Clinical Laboratory Evaluation | 32 |
| 4.15.4 | Vital Signs, Physical Findings and Other Observations Related to Safety | 33 |
| 4.15.5 | Other safety | 33 |
| 4.15.6 | Safety Monitoring (Independent Data Monitoring Committee [IDMC], Data | |
| | Monitoring Committee [DMC], Data and Safety Monitoring Board [DSMB]) | 33 |
| 4.16 | Determination of Sample Size | 34 |
| 4.17 | Changes in the Conduct of the Study or Planned Analysis | 34 |
| 5 | REFERENCES | 35 |
| 6 | Appendix | 36 |
| 6.1 | SAS program to reproduce data in Zhou et al [10]. | 36 |

Blue Earth Diagnostics BED-PSMA-301

Statistical Analysis Plan

## **REVISION HISTORY**

| Version No. | Effective Date | Summary of Change(s) |
|---|---|---|
| 1.0 | 03 July 2020 | Finalized document |
| 2.0 | 18 Aug 2021 | Added BMI |
| | _ | Wording: Replaced consensus between blinded readers with |
| | | majority of blinded readers. |
| | | Added that within analysis of subcategories, categories with |
| | | low counts may be collapsed. |
| | | Removed second exploratory objective and endpoint |
| | | Updated first exploratory endpoint to use cluster binary data |
| | | estimation of Confidence Interval |
| 3.0 | Date of Last | Changed TEAE definition from on or before Visit 3 to on or |
| | Signature | before Day 4. |
| | | Changed medications and/procedures starting after Day 4 not |
| | | to be summarized. |
| | | Changed summaries of TEAE leading to death, serious |
| | | adverse events, and discontinuation will only display TEAE. |

TP-GDO-WW-016-07.a CONFIDENTIAL **Project Document Version No.** 3.0 Effective Date: 30 Jan 19 **Project Document Effective Date**: Date of last signature Related to: SOP-GDO-WW-019 

Blue Earth Diagnostics BED-PSMA-301

Statistical Analysis Plan

## LIST OF ABBREVIATIONS

| Abbreviation / Acronym | Definition / Expansion |
|------------------------|----------------------------------------------|
| AE | Adverse event |
| BIE | blinded image evaluation |
| CI | Confidence interval |
| CSP | Clinical Study Protocol |
| COVID-19 | Coronavirus disease 2019 |
| CT CT | Computed tomography |
| DRM | Data Review Meeting |
| EBRT | External beam radiation therapy |
| EAP | Efficacy Analysis Population |
| ECG | electrocardiogram |
| eCRF | electronic Case Report Form |
| EEP | Extended Efficacy Population |
| FAS | Full Analysis Set |
| FN | False Negative |
| FP | False Positive |
| FSP | Full Safety Population |
| GGG | Gleason Grade Grouping |
| IP | Investigational product |
| IMP | Investigational Medicinal Product |
| IV | Intravenous |
| LN | Lymph Node |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MRI | Magnetic resonance imaging |
| NPV | Negative Predictive Value |
| PCa | Prostate Cancer |
| PET | Positron emission tomography |
| PLND | Pelvic lymph node dissection |
| PP | Per Protocol Population |

TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019 CONFIDENTIAL Project Document Version No. 3.0
Project Document Effective Date: Date of last signature


## Blue Earth Diagnostics

BED-PSMA-301 Statistical Analysis Plan

| Abbreviation / Acronym | Definition / Expansion |
|------------------------|----------------------------------|
| PPV | Positive predictive value |
| PSA | prostate-specific antigen |
| PT | Preferred Term |
| RP | Radical prostatectomy |
| SAE | Serious adverse event |
| SAP | Statistical Analysis Plan |
| SD | Standard Deviation |
| SOC | System Organ Class |
| SOP | Standard Operating Procedures |
| SoT | Standard of Truth |
| TEAE | Treatment-emergent adverse event |
| TLFs | Tables, Listings and Figures, |
| TN | True Negative |
| TP | True Positive |
| VDR | Verified Detection Rate |
| WHO-DD | WHO Drug Global |

TP-GDO-WW-016-07.a CONFIDENTIAL Project Document Version No. 3.0 Effective Date: 30 Jan 19 Project Document Effective Date: Date of last signature Related to: SOP-GDO-WW-019 

Blue Earth Diagnostics BED-PSMA-301

Statistical Analysis Plan

### 1 INTRODUCTION

Prostate cancer (PCa) is the most prevalent cancer in men in the developed world and the third leading cause of death (Jemal, 2011). It is most commonly diagnosed in men aged 65 years and over and in its early stages it is largely asymptomatic, with tumors detected by identification of increased levels of prostate-specific antigen (PSA) in peripheral blood. If detected early, and when the disease is organ confined, the 5-year survival rate approaches 100%.

Accurate staging of newly diagnosed PCa assists in directing appropriate treatment strategies. The National Comprehensive Cancer Network (NCCN Guidelines; Version 1.2020; PROS-2) recommend bone imaging and abdominal/pelvic imaging as the initial work-up in patients with newly-diagnosed high- and very high-risk PCa, as well as in a subgroup of patients with unfavorable intermediate-risk PCa. The primary goal of such imaging is to detect extra-prostatic disease (M1: non-regional nodal involvement, bone, or other sites [UICC, TNM Classification of Malignant Tumours]); the identification of which would likely significantly change the planned treatment regimen from locoregional to systemic therapy.

The overwhelming need for improved imaging should focus on the identification of N1 (metastasis in regional node(s)) and M1 disease, which may potentially have a meaningful impact on patient treatment and outcomes. Ideally, a staging technique that detects extra-prostatic disease should: 1) image the whole body, 2) not be limited to the skeleton, and 3) be both sensitive and specific for identifying PCa extent.

This study is designed to assess the performance of rhPSMA-7.3 (<sup>18</sup>F) for detecting N1 and M1 disease in patients with newly diagnosed PCa eligible for curative intent, standard of care locoregional therapy, who have elected to undergo radical prostatectomy (RP) with regional pelvic lymph node dissection (PLND). Evaluation of the sensitivity and specificity of rhPSMA-7.3 (<sup>18</sup>F) imaging by central blinded image evaluation (BIE) for detecting regional pelvic lymph node (LN) involvement, compared to histopathology, will be performed as the co-primary endpoints. Therefore, only patients who are scheduled to undergo RP and a PLND will be included in this study.

The Statistical Analysis Plan (SAP) details the statistical methodology to be used in analyzing study data and outlines the statistical programming specifications for the Tables, Listings and Figures (TLFs). It describes the variables and populations, anticipated data transformations and manipulations and other details of the analyses not provided in the Clinical Study Protocol (CSP). In case of discrepancies between Study Protocol and SAP the SAP supersedes the Study Protocol.

The SAP will be finalized prior to database lock and describes the statistical analysis as it is foreseen when the study is being planned. If circumstances should arise during the study rendering this analysis inappropriate, or if improved methods of analysis should arise, updates to the analyses may be made.

The analyses described in this SAP are based upon the following study documents:

- Study Protocol, Version 3.0 (July 01, 2020)
- Electronic Case Report Form (eCRF), Version 4.0 (February 8, 2021)

TP-GDO-WW-016-07.a CONFIDENTIAL **Project Document Version No.** 3.0 Effective Date: 30 Jan 19 **Project Document Effective Date**: Date of last signature Related to: SOP-GDO-WW-019 

Blue Earth Diagnostics BED-PSMA-301

Statistical Analysis Plan

- Invicro Independent Review Charter (IRC), Version 2.0 (June 18, 2021)
- Invicro Technical Operations Manual Version 4.0 (August 04, 2020)
- Invicro Review Session Methodology: Conventional Imaging Version 1.0 (June 08, 2021)

The following guidance document has been used:

Guidance for Industry and FDA Staff - Statistical Guidance on Reporting Results from Studies Evaluating Diagnostic Tests (13 March 2007)

### 2 STUDY OBJECTIVES

### 2.1 Primary Objective(s)

The primary objective of the study is to assess the sensitivity and specificity of rhPSMA-7.3 (<sup>18</sup>F) positron emission tomography (PET) in detecting N1 disease (as determined by the central BIE) on a patient level compared to the histopathology of pelvic lymphatic tissue removed during RP and PLND. At least one positive pelvic LN on PET (N1) and one positive LN as determined by histopathology (pN1) on the same side of the pelvis (left or right) will be deemed a True Positive (TP) at the patient level. In patients who have no TP regions (left or right), the translation of varying combinations of False Positive (FP), True Negative (TN) and False Negative (FN) regions to patient level categorizations is described in detail in Section 4.13.

## 2.2 Secondary Objective(s)

The secondary objectives of the study are:

- 1. To assess the Verified Detection Rate (VDR) for M1 disease of rhPSMA-7.3 (<sup>18</sup>F) PET findings (as determined by central BIE) on a patient level in patients with newly diagnosed unfavorable intermediate-, high-, or very high-risk PCa using histopathology or confirmatory imaging.
- 2. To assess the VDR for M1 disease of rhPSMA-7.3 (<sup>18</sup>F) PET findings (as determined by central BIE) on a patient level in patients with negative conventional imaging.
- 3. To assess the positive predictive value (PPV) of rhPSMA-7.3 (<sup>18</sup>F) PET for N1 and M1 lesions (as determined by central BIE) compared to histopathology or confirmatory imaging (M1 lesions only).
- 4. To assess the PPV of rhPSMA-7.3 (<sup>18</sup>F) PET for detecting pelvic LN metastases compared to surgical pathology on a patient level in which a FP patient is defined as having at least one FP region (right or left pelvis), regardless of any coexisting TP findings.
- 5. To assess the negative predictive value (NPV) of rhPSMA-7.3 (<sup>18</sup>F) PET for detecting pelvic LN metastases compared to surgical pathology on a patient level in which a FN patient is defined as having at least one FN region (right or left pelvis), regardless of any coexisting TN findings.
- 6. To assess the impact of rhPSMA-7.3 (<sup>18</sup>F) PET BIE on a) upstaging patients planned for RP or b) converting planned RP to external beam radiation therapy (EBRT).

TP-GDO-WW-016-07.a CONFIDENTIAL I Effective Date: 30 Jan 19 **Project Document E** Related to: SOP-GDO-WW-019

**Project Document Version No. 3.0** 

**Project Document Effective Date**: Date of last signature


Blue Earth Diagnostics BED-PSMA-301

Statistical Analysis Plan

- 7. To determine the inter- and intra-reader agreement of rhPSMA-7.3 (<sup>18</sup>F) scan interpretation by blinded independent readers.
- 8. To assess the safety of rhPSMA-7.3 (<sup>18</sup>F) injection in patients.

#### 2.3 **Exploratory Objective(s)**

The exploratory objectives of the study are:

1. To assess the sensitivity and specificity of rhPSMA-7.3 (<sup>18</sup>F) PET in detecting nodal metastases (as determined by central BIE) on a regional level compared to the histopathology of pelvic lymphatic tissue removed during RP and PLND.

### INVESTIGATIONAL PLAN

#### 3.1 **Overall Study Design and Plan**

This is a prospective, Phase 3, multi-center, single-arm, diagnostic imaging study designed to evaluate the safety and diagnostic performance of rhPSMA-7.3 (<sup>18</sup>F) PET ligand for the detection of N1 and M1 metastases in men with newly diagnosed unfavorable intermediate-, high- or very high-risk PCa (per NCCN Guidelines Version 1.2020; PROS-2).

Up to approximately 375 patients will be enrolled into the study to ensure inclusion of at least 300 evaluable patients undergoing RP and PLND. Consented patients will be screened at Visit 1 to determine eligibility for the study up to 28 days (up to 45 days due to the Coronavirus Disease-2019 [COVID-19] pandemic) before Investigational product (IP) administration at Visit 2. Due to the COVID-19 pandemic, Visit 1 and Visit 2 may be combined. Patients who meet all of the inclusion criteria and none of the exclusion criteria will be assigned a patient identifier (ID) and entered into the study at screening. In addition to their routine clinical work-up, which may include <sup>99m</sup>technetium-biphosphonate and abdominal/pelvic computed tomography (CT) or magnetic resonance imaging (MRI) and chest CT per local practice, and before the scheduled RP, patients will be administered a dose of rhPSMA-7.3 (<sup>18</sup>F), an administered activity of 8 mCi (296 MBq)  $\pm$  20% delivered as an intravenous (IV) bolus injection with a 10 mL fast 0.9% sodium chloride flush, followed by PET imaging.

Note: The screening/eligibility evaluation may take place on the day of rhPSMA-7.3 (<sup>18</sup>F) administration (with pre-screening via telephone), if necessary, to ensure the safety of enrolled patients (see Visit 1 and 2 combined; CSP Section 10.3). Alternatively, the time from Visit 1 (initial screening) to Visit 2 (rhPSMA-7.3 (<sup>18</sup>F) PET scan) may be extended to 45 days due to the COVID-19 pandemic.

The PET imaging results for each patient will be reported to the responsible physician prior to the planned RP. If safe and feasible, within 1 to 3 days post-IP administration, the patient must return to the clinic for safety follow-up including an electrocardiogram (ECG), blood safety laboratory tests and a focused physical examination. Clinical review of the imaging results and discussion of further procedures/treatments with the patient should also take place at this visit if the results are available. In cases where the rhPSMA-7.3 (<sup>18</sup>F) PET imaging results are not available at the safety

TP-GDO-WW-016-07.a CONFIDENTIAL **Project Document Version No. 3.0** Effective Date: 30 Jan 19 **Project Document Effective Date**: Date of last signature Related to: SOP-GDO-WW-019

Blue Earth Diagnostics BED-PSMA-301

Statistical Analysis Plan

follow-up visit, imaging results and further procedures/treatment plan should be discussed with the patient within 7 days after rhPSMA-7.3 (<sup>18</sup>F) imaging (this review may be conducted by telephone at the clinician's discretion). Note: due to the COVID-19 pandemic, the post-IP safety follow-up (laboratory and ECG assessments and focused physical examination) may be conducted within 1 to 5 days post-IP administration to ensure the safety of enrolled patients.

Within 45 days post-IP administration (may be extended to 60 days due to the COVID-19 pandemic), the patient will receive treatment as follows, with further detail provided in CSP Section 9.1.6.

- Standard of care surgical treatment of PCa, including a PLND; or
- If the rhPSMA-7.3 (<sup>18</sup>F) PET scan detects M1 lesion(s):
  - o A biopsy/surgery and/or additional imaging to confirm M1 lesion(s) will be required prior to initiation of treatment.

Safety will include adverse events (AEs) and vital signs monitoring, clinical laboratory evaluations, 12-lead ECG and focused physical examinations performed in all patients.

## 3.2 Endpoints

## 3.2.1 Primary Efficacy Endpoint

The co-primary endpoints for this study will be the:

- Sensitivity of rhPSMA-7.3 (<sup>18</sup>F) PET (as determined by central BIE) for detecting pelvic LN metastases compared to surgical pathology on a patient level.
- Specificity of rhPSMA-7.3 (<sup>18</sup>F) PET (as determined by central BIE) for detecting pelvic LN metastases compared to surgical pathology on a patient level

### 3.2.2 Secondary Efficacy Endpoints

The secondary endpoints for this study will be:

- 1. Percentage of patients in whom rhPSMA-7.3 (<sup>18</sup>F) imaging detects at least one verified M1 metastasis, as determined by central BIE.
- 2. Percentage of patients with negative conventional imaging for M1 disease in whom rhPSMA-7.3 (<sup>18</sup>F) PET detects at least one verified M1 metastasis, as determined by central BIE.
- 3. Patient level PPV of rhPSMA-7.3 (<sup>18</sup>F) PET BIE for N1 and M1 lesions compared to histopathology or confirmatory imaging (M1 lesions only).
- 4. PPV of rhPSMA-7.3 (<sup>18</sup>F) PET for detecting pelvic LN metastases compared to surgical pathology on a patient level in which a FP patient is defined as having at least one FP region (right or left pelvis), regardless of any coexisting TP findings.
- 5. NPV of rhPSMA-7.3 (<sup>18</sup>F) PET for detecting pelvic LN metastases compared to surgical pathology on a patient level in which a FN patient is defined as having at least one FN region (right or left pelvis), regardless of any coexisting TN findings.

6.

TP-GDO-WW-016-07.a CONFIDENTIAL **Project Document Version No.** 3.0 Effective Date: 30 Jan 19 **Project Document Effective Date**: Date of last signature Related to: SOP-GDO-WW-019 

Blue Earth Diagnostics BED-PSMA-301

Statistical Analysis Plan

- a. The percentage of patients being upstaged to N1 or M1 disease;
- b. The percentage of patients in whom planned RP is converted to EBRT.
- 7. Kappa statistic for the agreement between and within blinded independent readers on the interpretation of rhPSMA-7.3 (<sup>18</sup>F) scans.
- 8. Safety (AEs, vital signs clinical laboratory evaluations, 12-lead ECG and focused physical examinations) of rhPSMA-7.3 (<sup>18</sup>F) injection in patients

## 3.2.3 Exploratory Efficacy Endpoints

1. Diagnostic performance (sensitivity and specificity) of rhPSMA-7.3 (<sup>18</sup>F) PET for detecting pelvic LN metastases compared to surgical pathology on a regional level.

### 3.2.4 Safety Variables

In all patients, safety evaluations will include AE monitoring and reporting from the time of informed consent throughout the study.

Vital sign assessments will also be conducted at screening and pre- and post-IP administration on the day of rhPSMA-7.3 (<sup>18</sup>F) injection.

In addition, a focused physical examination will be performed at screening and at the safety follow-up visit within 1 to 3 days post-IP administration (may occur within 1 to 5 days post-IP administration due to the COVID-19 pandemic), and a 12-lead ECG will be performed pre-IP administration on the day of rhPSMA-7.3 (<sup>18</sup>F) injection and at the safety follow-up visit within 1 to 3 days post-IP administration (may occur within 1 to 5 days post-IP administration due to the COVID-19 pandemic). Baseline blood safety laboratory tests, including hematology (full blood count), biochemistry (urea and electrolytes, liver function tests) and coagulation will be performed pre-IP administration on the day of rhPSMA-7.3 (<sup>18</sup>F) injection and repeated at the safety follow-up visit within 1 to 3 days post-IP administration (may occur within 1 to 5 days post-IP administration due to the COVID-19 pandemic).

### 4 STATISTICAL METHODS

### 4.1 Data Quality Assurance

All tables, figures and data listings to be included in the report will be independently checked for consistency, integrity and in accordance with standard Parexel procedures.

### 4.2 General Presentation Considerations

'Baseline' is defined as the last available pre-IP administration assessment.

'End of Study' is defined as the last available post-IP administration assessment.

TP-GDO-WW-016-07.a CONFIDENTIAL **Project Document Version No.** 3.0 Effective Date: 30 Jan 19 **Project Document Effective Date**: Date of last signature Related to: SOP-GDO-WW-019 

Blue Earth Diagnostics BED-PSMA-301

Statistical Analysis Plan

- 'Study Day' will be calculated relative to the date of rhPSMA\_7.3 (<sup>18</sup>F) injection day, and is equal to:
  - Assessment Date IP Administration Date + 1 if the assessment date is on or after IP administration date.
  - <u>Assessment Date IP Administration Date, if the assessment date is before IP administration date.</u>

Continuous data will be summarized in terms of the mean, standard deviation (SD), median, minimum, maximum and number of observations, unless otherwise stated. Continuous data (e.g. counts) that are expected to be skewed will be presented in terms of the maximum, upper quartile, median, lower quartile, minimum and number of observations. The minimum and maximum will be reported to the same number of decimal places as the raw data recorded in the database. The mean, median, lower quartile and upper quartile will be reported to one more decimal place than the raw data recorded in the database. The SD will be reported to two more decimal places than the raw data recorded in the database. In case the rules result in more than four decimal places, the number of decimal places reported shall be four for any summary statistic, irrespective of the previous rules.

Categorical data will be summarized in terms of the number of patients providing data at the relevant time point (n), frequency counts and percentages. Any planned collapsing of categories will be detailed in the SAP text and the data displays.

Percentages will be presented to one decimal place. Percentages will not be presented for zero counts. Percentages will be calculated using n as the denominator. If sample sizes are small, the data displays will show the percentages, but any textual report will describe frequencies only.

Changes from baseline in categorical data will be summarized using shift tables where appropriate.

P-values greater than or equal to 0.001, in general, will be presented to three decimal places. P-values less than 0.001 will be presented as "<0.001".

Confidence intervals (CIs) of continuous variables will be presented to one more decimal place than the raw data. CIs of proportions will be presented to three decimal places (e.g. 1/3 will be a proportion of 0.333) and exact intervals (Clopper-Pearson) will be employed unless specified otherwise. CI for percentages will be to one decimal place.

### 4.3 Software

All report outputs will be produced using SAS® version 9.3 or a later version in a secure and validated environment.

TP-GDO-WW-016-07.a CONFIDENTIAL Project Document Version No. 3.0 Effective Date: 30 Jan 19 Project Document Effective Date: Date of last signature Related to: SOP-GDO-WW-019 

Blue Earth Diagnostics BED-PSMA-301

Statistical Analysis Plan

## 4.4 Study Patients

### 4.4.1 Disposition of Patients

A clear accounting of the disposition of all patients who enter the study will be provided, from screening to study completion as per CONSORT guidance.

The following summaries will be provided:

- A summary of the number of patients screened for entry into the study and the number and percentage of patients excluded prior to IP administration by major reason and overall (Analysis set: All enrolled Patients)
- A summary of the number of patients enrolled (See section 4.5) per center, and per country (Analysis set: Full Analysis Set [FAS]).
- A summary of the number of patients who received IP, number of patients who had an evaluable PET scan following IP administration, and the number and percentage of patients withdrawing from the study and completing each phase. (Analysis set: FAS).
- A summary of withdrawals from the study and from IP administration by major reason (Analysis set: FAS).

By-patient listings of eligibility details, enrollment details, visit dates (including impact of COVID-19 on visits), withdrawal/study completion details (including reason for discontinuation and time since IP administration prior to discontinuation) will be provided.

### 4.4.2 Protocol Deviations

Protocol deviations will be handled in accordance with Parexel Standard Operating Procedures (SOPs).

Protocol deviations occur when the patient, investigator, or Sponsor fails to adhere to protocol requirements or where there is a significant non-compliance to ICH-GCP, affecting patient safety or the scientific value of the trial.

Major protocol deviations are defined as those deviations from the protocol likely to have an impact on the perceived efficacy and/or safety of study treatments. The impact of major protocol deviations on the efficacy and/or safety results will be investigated by assessing the robustness of the study results and conclusions to the choice of analysis set, both including and excluding data potentially affected by major protocol deviations at a Data Review Meeting (DRM) shortly before database lock. Results and population assignments will be summarized in a DRM report which will be signed off by all relevant scientific experts.

Major protocol deviations and any action to be taken regarding the exclusion of patients or affected data from specific analyses are defined in the project-specific Protocol Deviation Specification which is agreed and signed off before analysis.

Major protocol deviations which lead to withdrawal and replacement of the patient include, but not limited to:

TP-GDO-WW-016-07.a CONFIDENTIAL Project Document Version No. 3.0 Effective Date: 30 Jan 19 Project Document Effective Date: Date of last signature Related to: SOP-GDO-WW-019 

Blue Earth Diagnostics BED-PSMA-301

Statistical Analysis Plan

- Failure to meet inclusion/exclusion criteria (see CSP Sections 6.2 and 6.3).
- Use of a prohibited concomitant medication (see CSP Section 7.1).
- IP administration but no subsequent PET scan.
- Significant non-compliance with IP administration.

Patients will be withdrawn from the study and be included in the All Enrolled Patients and Full Safety Population as applicable.

Deviations due to COVID-19 will be listed separately.

A by-patient listing of major protocol deviations will be provided.

A summary of the number and percentage of patients with a major protocol deviation by type of deviation (Analysis set: FAS) will be provided.

## 4.5 Analysis Sets

All enrolled patients: all patients who signed the informed consent form.

Full Analysis Set (FAS): all patients who were scheduled to receive the rhPSMA-7.3 (<sup>18</sup>F) injection having met the inclusion/exclusion criteria.

Full Safety Population (FSP): all patients who received the rhPSMA-7.3 (<sup>18</sup>F) injection.

**Efficacy Analysis Population (EAP):** all patients who received rhPSMA-7.3 (<sup>18</sup>F) injection followed by a PET/CT scan and who underwent RP and PLND.

**Extended Efficacy Population (EEP):** all patients who received rhPSMA-7.3 (<sup>18</sup>F) injection followed by a PET/CT scan. This population includes M0 and M1 patients independent of performance of RP and PLND and will be used for M1 related efficacy and Kappa statistics.

**Per Protocol Population (PP):** All patients in the EAP population who have histology available from surgery that allows SoT determination, and without any major protocol deviations that will affect the evaluations of the PET scan or histology.

The primary analysis will be based on the EAP. The FSP will be used for all safety summaries.

Upon database release, protocol deviation and analysis set outputs will be produced and will be to BED for review. An analysis set classification meeting will be arranged to discuss the outputs and to decide which patients and/or patient data will be excluded from certain analyses. Decisions made regarding the exclusion of patients and/or patient data from the analyses, and the agreement of population inclusion for each patient, will be made prior to database lock and will be documented and approved by the Sponsor.

A by-patient listing of analysis set details will be provided. This listing will include: center, country, patient identifier, and inclusion/exclusion flag for each set and reason for exclusion from

TP-GDO-WW-016-07.a CONFIDENTIAL
Effective Date: 30 Jan 19 Project Docume
Related to: SOP-GDO-WW-019

**Project Document Version No. 3.0** 

**Project Document Effective Date**: Date of last signature


Blue Earth Diagnostics BED-PSMA-301

Statistical Analysis Plan

each set. All enrolled patients will appear on this listing. If patient data have been partially excluded, visit will also appear on this listing.

The number and percentage of patients in each population will be provided using all enrolled patients.

### 4.6 Demographic and Other Baseline Characteristics

## 4.6.1 Demographics

All demographics (e.g. age [including age groups of  $<65, \ge65$  and the subgroup of  $\ge75$ ], sex, race, height, weight and BMI at screening and on Day 1) and baseline characteristics will be listed, and their baseline characteristics summarized (with weight and BMI on day 1) using the FAS, FSP, EAP, EEP and PP.

BMI will be calculated as 
$$BMI(kg/m^2) = \frac{weight(kg)}{height(m)^2}$$

### 4.6.2 Baseline conventional imaging

Baseline conventional imaging will be taken from imaging performed within the 60 days before screening or will be performed prior to IP administration.

The imaging results classified as baseline (above) will be summarized using FAS, EAP, EEP and PP by imaging modality and as positive or negative for detection of N1 or M1 disease. Patients with more than one baseline scan will be summarized for the combination of baseline scans and include all applicable anatomical areas covered. A listing will contain all these baseline parameters and include the imaging modality (CT, MRI, bone Scan, etc).

### 4.6.3 Prostate Cancer History

Prostate cancer history will be summarized using the FAS, FSP, EAP, EEP and PP for time of initial prostate cancer diagnosis to informed consent (in months), for TNM stage, total Gleason score (Frequencies), Gleason Grade Group (GGG) based on prostate biopsy, most recent PSA including frequency by categorization (0-0.5, >0.5-1.0, >1.0-2.0, >2.0-5.0, >5.0-10.0, >10.0 [ug/L]).

This same information will be listed by patient.

Gleason Grade Group is defined by the International Society of Urological Pathologists, and the categories are as follows:

- Grade Group 1 is defined as Total Gleason score ≤6
- Grade Group 2 is defined as Gleason score 3+4=7
- Grade Group 3 is defined as Gleason score 4+3=7
- Grade Group 4 is defined as Total Gleason score of 8
- Grade Group 5 is defined as Total Gleason scores 9-10

TP-GDO-WW-016-07.a CONFIDENTIAL **Project Document Version No.** 3.0 Effective Date: 30 Jan 19 **Project Document Effective Date**: Date of last signature Related to: SOP-GDO-WW-019 

Blue Earth Diagnostics BED-PSMA-301

Statistical Analysis Plan

TNM staging will be displayed at observed level and combined at levels T2, T3, T4, M0, M1, MX, where each of these contain underlying categories (i.e. T2 -All contains subjects with observed at T2, T2a, T2b, T2c)

### 4.6.4 Baseline Risk Category

Risk Category will be assigned using the NCCN Guidelines, version 1.2020; PROS-2. A listing of risk category and underlying variables will be provided. Risk category will be summarized into categories using the EAP. Risk Categories are shown in Table 1. Per the CSP, risk categories of unfavorable intermediate-risk, high-risk or very high-risk are expected.

Table 1: Risk Categories from NCCN guidelines.

| Risk Group | Clinical/Pathologic Features |
|---|---|
| Very Low | T1c AND |
| | Grade Group 1 AND |
| | PSA <10 ng/mL AND |
| | Fewer than 3 prostate biopsy fragments/cores positive, ≤50% cancer in each fragment/core AND |
| | PSA density < 0.15 ng/mL/g |
| Low | Has all following but does not qualify for very low risk |
| | T1-T2a AND |
| | Grade Group 1 AND |
| | PSA < 10 ng/mL |
| Favorable | No High or Very High-risk features |
| intermediate | 1 Intermediate Risk Factors and |
| | Grade Group 1 or 2 and |
| | <50% biopsy cores positive |
| Unfavorable | No High or Very High-risk features |
| Intermediate | 2 or 3 Intermediate Risk Factors. and/or |
| | Grade Group 3 and/or |
| | ≥50% biopsy cores positive |
| High | No very-high risk features and has at least one high-risk feature: |
| | T3a OR |
| | Grade Group 4 or Grade Group 5 OR |
| | PSA>20 ng/mL |
| Very High | Has at least one of the following |
| | T3b-T4 OR |
| | Primary Gleason pattern 5 OR |
| | 2 or 3 high-risk features |
| | >4 cores with Grade Group 4 or 5 |

Intermediate risk factors are: T2b-T2c, PSA 10-20 ng/mL, Grade Group 2 or 3

In this study, the risk groups will be categorized into:

- "High or Very High Risk" defined as meeting any one of these criteria: T-stage T3 (including T3a and T3b) or T4, Gleason Grade Group 4 or 5, Primary Gleason pattern 5, or PSA >20ng/mL
- "Not High or Very High Risk" defined as not meeting any of the criteria meeting the high or very high-risk criteria.

TP-GDO-WW-016-07.a CONFIDENTIAL Project Document Version No. 3.0 Effective Date: 30 Jan 19 Project Document Effective Date: Date of last signature Related to: SOP-GDO-WW-019 

Blue Earth Diagnostics BED-PSMA-301

Statistical Analysis Plan

## 4.6.5 Medical history

Medical history will be coded using Medical Dictionary for Regulatory Activities (MedDRA) version 22.1 or higher – the data will be listed and include start date, end date, ongoing at study start, Preferred Term (PT) and System Organ Class (SOC). Medical history will also be summarized using FSP by SOC and PT.

### 4.7 Prior and Concomitant Medications and Procedures

Medication and/or procedure start and stop dates will be compared to the date of IP administration to allow medications/procedures to be classified as either Prior only, both Prior and Concomitant, or Concomitant only. Medications and/or procedures starting after Day 4 will be listed but will not be classified or summarized.

Medications/procedures that start and stop prior to the date of dose of IP administration will be classified as Prior only. If a medication/procedure starts before the date of IP administration and stops on or after the date of IP administration, then the medication/procedure will be classified as both Prior and Concomitant. Medications/procedures will be classified as Concomitant only if they have a start date on or after the date of first dose of study medication.

If medication/procedure start and/or stop dates are missing or partial, the dates will be compared as far as possible with the date of IP administration. Medications/procedures will be assumed to be Concomitant only, unless there is clear evidence (through comparison of partial dates) to suggest that the medication/procedure started prior to the IP administration. If there is clear evidence to suggest that the medication/procedure started prior to the IP administration, the medication/procedure will be assumed to be both Prior and Concomitant, unless there is clear evidence to suggest that the medication/procedure stopped prior to the IP administration. If there is clear evidence to suggest that the medication/procedure stopped prior to the IP administration, the medication will be assumed to be Prior only.

Medications will be coded using WHODrug Global Dictionary and summarized by ATC code (levels 2 and 4) and Preferred term and listed by patient using the FSP. In case of missing level 4 coding the level 3 coding will be used.

Procedures will be summarized by System Organ Class (SOC) and Preferred Term (PT) using MedDRA dictionary and listed by patient.

All prior and concomitant medications and procedures will be listed by patient. Concomitant medications will be summarized using the FSP.

### 4.8 Exposure and Treatment Compliance

A patient listing of rhPSMA-7.3 (<sup>18</sup>F) administration including total administered activity, injection site reactions, local imaging results, incidental findings, and evaluations of the independent blinded central PET readers will be provided.

TP-GDO-WW-016-07.a CONFIDENTIAL **Project Document Version No.** 3.0 Effective Date: 30 Jan 19 **Project Document Effective Date**: Date of last signature Related to: SOP-GDO-WW-019 

Blue Earth Diagnostics BED-PSMA-301

Statistical Analysis Plan

A summary of total administered activity will be provided using the FAS and PP. All activity will be converted to MBq using the conversion 1mCi=37 MBq.

## 4.9 rhPSMA-7.3 (<sup>18</sup>F) Image reading

Each rhPSMA-7.3 (<sup>18</sup>F) image will initially be read by a site-based local reader, and the results will be listed including incidental findings. In addition, for the primary endpoint analysis, imaging will be read by three blinded independent PET readers (see the study Independent Review Charter for further details). The results of the blinded PET readers will be used in the primary analysis, thus requiring each (statistical) analysis to be performed three times. In addition, the majority interpretation will be displayed.

Table 2 Derivation of Overall Interpretation (2 out of 3 readers consensus)

| Reader 1 | Reader 2 | Reader 3 | Majority |
|----------|----------|----------|----------|
| Positive | Positive | Positive | Positive |
| Positive | Positive | Negative | Positive |
| Negative | Negative | Positive | Negative |
| Negative | Negative | Negative | Negative |

PET imaging results (i.e. positive/negative) will be summarized using the EEP by anatomical location by category and anatomical location within category. Categories will be prostate, pelvic lymph nodes, lymph nodes outside of pelvis, soft tissue/parenchyma and bones, as well as extrapelvic (which would include lymph nodes outside of pelvis, soft tissue/parenchyma and bones together). All categories will be presented in the summary, but anatomical locations will only be presented where data are collected, i.e. lesion investigated in that anatomical location.

### 4.10 Biopsy/Surgery

If the rhPSMA-7.3 (<sup>18</sup>F) PET shows M1 metastatic disease, the patient will be asked to undergo a biopsy or confirmatory imaging of the PET-positive lesion(s) to confirm the presence of a metastasis. If a surgical intervention of this lesion is carried out as part of the treatment, this may substitute for a biopsy. If the patient has proven M1 metastatic disease, the disease management may be altered, based on the responsible physician's clinical judgement. This change in disease management will be documented on the eCRF.

If rhPSMA-7.3 (<sup>18</sup>F) PET does not detect M1 disease, the patient will undergo the scheduled RP and PLND. In patients without M1 lesions identified and in whom the patient and physician believe, after obtaining the results of the rhPSMA-7.3 (<sup>18</sup>F) PET, that EBRT would be a better therapeutic option than surgery, the patient may proceed to EBRT and the rationale for this change of disease management will be documented on the eCRF.

TP-GDO-WW-016-07.a CONFIDENTIAL Project Document Version No. 3.0 Effective Date: 30 Jan 19 Project Document Effective Date: Date of last signature Related to: SOP-GDO-WW-019 

Blue Earth Diagnostics BED-PSMA-301

Statistical Analysis Plan

The regional PLND must be performed by a suitably qualified surgeon and should include, at minimum, resection of lymphatic tissue for histological analysis from the following nodal groups: 1) hypogastric (internal iliac), 2) external iliac, and 3) obturator LNs. Extended LN dissection may be performed if clinically appropriate and the anatomical regions (e.g. presacral, common iliac, peri-rectal) with left/right designations, should be recorded on the eCRF. The location of the dissected material shall be marked in order to allow matching with their anatomical origin (left and right pelvis); the left and the right side of the specimen shall be clearly marked. The dissected LNs will be sectioned and analyzed by a pathologist for the presence or absence of PCa according to standard of care at the clinical site. The number of lymph nodes sampled and found positive for PCa will be registered and summarized.

Patients with PET M1 will be summarized using the EEP by confirmatory method(s), result of confirmation, change in disease management, surgery (radical prostatectomy and pelvic lymph node dissection) performed, Lymph node dissection and (additional) treatment received. All counts will be presented including percentage of patients categorized as PET M1.

Patients will be summarized using the EEP by surgery (RP and PLND) received, extended lymph node dissection and (additional) treatment received. All counts will be presented including the percentage of patients categorized as PET M0.

Results by patient will be listed for both M0 and M1 patients. A display of Histopathology of Pelvic Lymph Nodes and a display of confirmatory procedures will be created for all patients. For M1 patients, a listing of PSMA Positive M1 Lesions (by anatomic location), including method (Biopsy/histopathology, CT Scan, MRI, Bone scan, Other) and result, will be created. A summary will be provided on methods to obtain standard of truth.

### 4.11 TNM staging and Gleason score

In addition to baseline values (Section 4.6.3), baseline and post-surgery staging will be summarized for TNM stage, primary and secondary and total Gleason score similar to baseline using the EEP. In addition, for GGG, a shift table will be presented from baseline to final staging.

### 4.12 Standard of Truth

Histology or confirmatory imaging will be used as the Standard of Truth (SoT), as defined below.

- 1. Histology
  - a. Histology of surgically removed pelvic LNs;
  - b. Histology obtained by biopsy of M1 lesion.
- 2. Confirmatory Imaging
  - a. In patients without available histopathology, confirmatory conventional imaging is acceptable as proof of M1 disease in case of unequivocal findings (e.g. sclerotic bone lesions on CT, positive bone lesions on bone scan, evidently enlarged LNs radiologically considered metastases, lesions in the liver representing metastases as determined by ultrasound, CT or MRI, multiple pulmonary nodules on CT).

TP-GDO-WW-016-07.a CONFIDENTIAL **Project Document Version No.** 3.0 Effective Date: 30 Jan 19 **Project Document Effective Date**: Date of last signature Related to: SOP-GDO-WW-019 

Blue Earth Diagnostics BED-PSMA-301

Statistical Analysis Plan

- b. Confirmatory imaging for proof of M1 disease will be read centrally. Three central reviewers will review all submitted imaging and reach consensus on the nature of the target lesion. Reads of the confirmatory imaging as SoT will be directed by rhPSMA-7.3 (<sup>18</sup>F) PET findings (for confirmation of lesion location only). A brief summary of clinical information will be available to the SoT readers (e.g. 67-year-old male with newly diagnosed, localized prostate cancer prior to rhPSMA-7.3 (<sup>18</sup>F) scan). Readers will be blinded to all other information. Further details are given in the study Independent Review Charter.
- 3. Baseline Conventional Imaging only
  - a. If M1 lesion identified by blinded PET reader but not site reader, or if M1 lesion is identified by site reader but no histology or no confirmatory imaging is available, then only conventional imaging at baseline will be used to determine the SoT.

SoT will be listed next to the results of the blinded independent reads and include method (Histology/Confirmatory Imaging/Baseline Imaging only), anatomical location and Result(s) using the EEP. Histology SoT will be assessed based on local reads of the PET scan, and these results will be included irrespective of BIE reading. The SoT will be summarized by method and anatomical location.

### 4.13 Hemipelvis Region Categorization and Patient Level Categorization

At least one positive pelvic LN on PET (N1) and one positive LN as determined by histopathology (pN1) on the same side of the pelvis (left or right), as depicted in Table 3, will be deemed a TP on a patient level.

**Table 3 Hemipelvis Region Categorization Method** 

| | At Least One Pathology-positive LN in the Region | No Pathology-positive LN in the Region |
|---|---|---|
| At Least One PET-Positive LN in the Region | True Positive (TP) region | False Positive (FP) region |
| No PET-positive LN in the Region | False Negative (FN) region | True Negative (TN) region |

LN=lymph node; PET=positron emission tomography.

For patients who have no TP regions, Table 4 depicts the method for assigning patient level categorizations based on by-region results (i.e. for the different possible hemipelvis combinations of TN, FN and FP regions).

Two analyses will be performed based on the classification of patients with one positive region and one negative region. The primary analysis will include patients as FN if they only had one positive region by histopathology and it was missed by PET. Full diagnostic statistics will be provided for both patient level classifications.

TP-GDO-WW-016-07.a CONFIDENTIAL Project Document Version No. 3.0 Effective Date: 30 Jan 19 Project Document Effective Date: Date of last signature Related to: SOP-GDO-WW-019 

Blue Earth Diagnostics BED-PSMA-301

Statistical Analysis Plan

### Table 4: Translation of Region Level to Patient Level Categorizations in Patients with No TP Regions

a)

| Patient Level Categorization | At Least one True<br>Negative (TN)<br>Region | At Least one False<br>Negative (FN) Region | At Least one False<br>Positive (FP) Region |
|---|---|---|---|
| True Negative (TN) | Yes | No | No |
| False Negative (FN) | Yes | Yes | No |
| False Negative (FN) | No | Yes | No |
| False Positive (FP) | Yes | No | Yes |
| False Positive (FP) | No | No | Yes |
| False Negative (FN) for Primary<br>Analysis; False Positive (FP) for<br>Secondary Analysis* | No | Yes | Yes |

PPV=positive predictive value.

b)

| Histopathology | PET Patient Level Classification | | | |
|---|---|---|---|---|
| | True Positive (TP) | False Negative (FN) | False Positive (FP) | True Negative<br>(TN) |
| Two Positive<br>Regions | 1 or 2 positive<br>regions on PET | Both regions negative on PET | NA | NA |
| One Positive<br>Region; One<br>Negative<br>Region | PET is correct on positive region | Primary analysis: PET is negative on the positive region Secondary analysis: PET is negative on both | Primary analysis: NA Secondary analysis: PET is negative on histopathology | NA |
| | | regions only | positive region and PET is<br>positive on histopathology<br>negative region | |
| Two Negative<br>Regions | NA | NA | PET-positive on one or two regions | PET is negative on both regions |

NA=cell classification is not applicable; PET=positron emission tomography.

Results of the Hemipelvis Categorization will be listed by region and summarized by region status using the EAP. This summary will include a category for missing Hemipelvis Categorization. The patient's by region and patient level classification will be listed including classification for the secondary analysis (Section 4.14.3.4 and 4.14.3.5).

A cross table of patients PET image diagnostic and SoT diagnostic will be provided.

TP-GDO-WW-016-07.a CONFIDENTIAL **Project Document Version No.** 3.0 Effective Date: 30 Jan 19 **Project Document Effective Date**: Date of last signature Related to: SOP-GDO-WW-019 

<sup>\*</sup> Patient contributes to the primary efficacy analysis for Sensitivity (False Negative categorization) and a secondary analysis of PPV (False Positive categorization).

Blue Earth Diagnostics BED-PSMA-301

Statistical Analysis Plan

## 4.14 Efficacy Evaluation

Unless otherwise stated, all efficacy evaluations will be done using the EAP as defined in Section 4.5.

### 4.14.1 Analysis and Data Conventions

The primary hypothesis involves a joint assessment of sensitivity and specificity against individual performance goals:

H<sub>0</sub>: Sensitivity  $\leq$  Se<sub>0</sub> or Specificity  $\leq$  Sp<sub>0</sub> versus H<sub>1</sub>: Sensitivity > Se<sub>0</sub> and Specificity > Sp<sub>0</sub> Where Se<sub>0</sub> and Sp<sub>0</sub> are performance goals for sensitivity and specificity, respectively. Performance goals of 22.5% (Se<sub>0</sub>) for sensitivity and 82.5% (Sp<sub>0</sub>) were selected based on the low sensitivity but high specificity of other PSMA ligands used for lymph node staging.

The definition of Sensitivity will be:

True Positive / (True Positive + False Negative)

The definition of Specificity will be:

True Negative / (True Negative + False Positive)

Additional analysis will be performed for PPV and NPV.

The definition of PPV will be:

True Positive / (True Positive + False Positive)

The definition of NPV will be:

True Negative / (True Negative + False Negative)

The sensitivity, specificity, PPV and NPV, together with the corresponding 95% CIs, will be estimated for each of the three blinded PET readers. All analyses performed for the three blinded PET readers will be repeated for their majority evaluation (Section 4.9).

# 4.14.1.1 Adjustments for Covariates

Not applicable.

### 4.14.1.2 Handling of Dropouts or Missing Data

Missing evaluation results in the biopsy/surgery will be assigned the worst value. Hence, a side with a positive rhPSMA-7.3 (<sup>18</sup>F) PET will be considered as false positive (i.e. SoT will be set to negative), while a side with negative rhPSMA-7.3 (<sup>18</sup>F) PET will be a false negative (i.e. SoT set to positive).

The number and percentage of patients with missing data for the biopsy/surgery will be summarized by major reason, as indicated in Section 4.13.

Imputation of missing dates for concomitant medications and procedures is described in Section 4.7, imputation of missing dates for AEs is described in Section 4.15.1.

TP-GDO-WW-016-07.a CONFIDENTIAL Project Document Version No. 3.0 Effective Date: 30 Jan 19 Project Document Effective Date: Date of last signature Related to: SOP-GDO-WW-019 

Blue Earth Diagnostics BED-PSMA-301

Statistical Analysis Plan

## 4.14.1.3 Interim Analyses

Using the first 150 patients an interim analysis of safety data will be created. The actual outputs for this are indicated in the shells.

### 4.14.1.4 Examination of Subgroups

The attributes of the primary efficacy variable will be examined across subgroups based on:

- PCa risk categories (high- or very high-risk vs not high or very high risk).
- Most recent PSA values (0-0.5, >0.5-1.0, >1.0-2.0, >2.0-5.0, >5.0-10.0, >10.0 [ng/mL])
- Race (Black or African American, American Indian or Alaska Native, Asian, Native Hawaiian or Other Pacific Islander, White, Not Reported, Other)
- Age (<65,>=65 and >=75)

The analysis within subgroups will involve the confidence intervals (CI) but not the hypothesis testing. For each of these analyses, if a category has low counts (less than 10) it may be collapsed with another category, for ordinal parameters only with neighboring categories.

A cross table of N1 disease status from rhPSMA-7.3 (<sup>18</sup>F) PET against to histopathology of pelvic LNs will be provided by risk category and associated 95% CI for Sensitivity and Specificity will be presented.

### 4.14.1.5 Clustered binary data estimate of variance

### 4.14.1.5.1 Sensitivity

Following Zhou et al. the following estimators will be used:

$$\widehat{Se} = \sum_{i=1}^{I} N_i * \widehat{Se}_i / \sum_{i=1}^{I} N_i$$

$$\widehat{Var}(\widehat{Se}) = \frac{1}{I(I-1)} \sum_{i=1}^{I} \left[ \frac{N_i}{\overline{N}} (\widehat{Se}_i - \widehat{Se})^2 \right]$$

With:

Se : Sensitivity

i : individual patient

I : total number of patients

N<sub>i</sub>: Number of elements (True Positive + False Negative) for patient i

 $\widehat{Se}_i$  : Sensitivity for patient i : Mean cluster size

The example in Zhou et al. is coded in SAS in Appendix 6.1.

An asymptotic normal distribution for the sampling distribution of  $\widehat{PPV}$  is assumed and the 95% confidence interval will be derived as:

$$\widehat{Se} \pm Z_{1-\alpha/2} \sqrt{\widehat{Var}(\widehat{Se})}$$

where  $Z_{1-\alpha/2}$  is the upper 1- $\alpha/2$  value for the standard normal distribution.

TP-GDO-WW-016-07.a CONFIDENTIAL **Project Document Version No.** 3.0 Effective Date: 30 Jan 19 **Project Document Effective Date**: Date of last signature Related to: SOP-GDO-WW-019 

Blue Earth Diagnostics BED-PSMA-301

Statistical Analysis Plan

## 4.14.1.5.2 Additional Confidence interval Sensitivity

Normal approximation in constructing 95% CIs might lead to bounds exceed [0, 1] for  $\widehat{PPV}$ . Hence an additional CI will be derived. Logit transformation will be applied to PPV and Delta Method (Casella and Berger, 2021) will be utilized to obtain to approximate the variance of logit(PPV). Accordingly, the asymptotical distribution of logit(PPV) is

$$\sqrt{n} \left[ log \left( \frac{\widehat{Se}}{1 - \widehat{Se}} \right) - log \left( \frac{Se}{1 - Se} \right) \right] \stackrel{d}{\to} N \left( 0, \frac{1}{[Se(1 - Se)]^2} Var \left( Se \right) \right).$$

Accordingly, an asymptotic normal distribution for the sampling distribution of  $logit(\widehat{Se})$  is assumed and the 95% confidence interval will be derived as:

$$logit(\widehat{Se}) \pm Z_{1-\alpha/2} \sqrt{\widehat{Var}(logit(\widehat{Se}))}$$

where  $Z_{1-\alpha/2}$  is the upper  $1-\alpha/2$  value for the standard normal distribution and  $\sqrt{\widehat{Var}(logit(\widehat{Se}))} \approx \frac{1}{[\widehat{Se}(1-\widehat{Se})]^2}\widehat{Var}(\widehat{Se})$ . Lower and upper confidence intervals values will be reported in [0,1] scale by the logit inverse transformation, as follows

$$CI_{[0,1]\,scale} = \frac{e^{CI\_logit}}{1 + e^{CI\_logit}}$$

## 4.14.1.5.3 Specificity

The formulas for sensitivity can be used with appropriate substitution.

Sensitivity=True Positive / (True Positive + False Negative)

Specificity=True Negative / (True Negative + False Positive)

### 4.14.2 Primary Efficacy Variable

The co-primary endpoints for the study are based on the sensitivity and specificity of rhPSMA-7.3 (<sup>18</sup>F) PET (by central BIE) in detecting N1 disease compared to histopathology of pelvic LNs. The primary analysis involves a joint assessment of sensitivity and specificity against individual performance goals:

## H<sub>0</sub>: Sensitivity $\leq$ Se<sub>0</sub> or Specificity $\leq$ Sp<sub>0</sub> versus H<sub>1</sub>: Sensitivity > Se<sub>0</sub> and Specificity > Sp<sub>0</sub>

Where  $Se_0$  and  $Sp_0$  are performance goals for sensitivity and specificity, respectively. Performance goals of 22.5% ( $Se_0$ ) for sensitivity and 82.5% ( $Sp_0$ ) for specificity were selected based on the low sensitivity but high specificity of other PSMA ligands used for LN staging. The analyses for sensitivity and specificity will be performed using one-sided 0.025 exact binomial tests. In addition to the rates, exact two-sided 95% CIs will also be provided. If the predefined sensitivity and specificity goals are met by the same two of three blinded independent readers (both tests reach statistical significance [P<0.05] for the same two readers), the study will be considered to have successfully demonstrated the effectiveness of the rhPSMA-7.3 ( $^{18}F$ ) in detecting N1 disease.

The TP, FP, TN and FN regions will be categorized according to Table 3 (Section 4.13) using a right and left hemipelvis regional classification method. For the primary analysis, patients who have one TP region will be categorized as a TP patient.

TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019 CONFIDENTIAL Project Document Version No. 3.0

Project Document Effective Date: Date of last signature

**Project Document Effective Date**: Date of last signature


Blue Earth Diagnostics BED-PSMA-301

Statistical Analysis Plan

For patients who have no TP regions, Table 4 depicts the method for assigning patient level categorizations based on by-region results (i.e. for the different possible hemipelvis combinations of TN, FN and FP regions).

Classification will be summarized via a cross table of region status using the layout of Table 4b. A summary of frequency of PET Patient level Classifications will be supplied including estimates and CI of Sensitivity and Specificity according to each blinded reader. Sensitivity and Specificity will be plotted for each reader including CI and performance goals.

The primary analysis will be repeated using the PP following methods of the primary analysis: A summary of frequency of PET Patient level Classifications will be supplied including estimates and CI of Sensitivity and Specificity according to each blinded reader. Frequencies will be displayed in a bar chart. Sensitivity and Specificity will be plotted for each reader including CI and performance goals.

### 4.14.2.1 Sensitivity Analysis; patients with FN and FP results

The primary efficacy analysis will be repeated with a reclassification of patients with one FN and one FP region. In particular, in the sensitivity analysis, these patients will be classified as FN. The results will be displayed in a summary of frequency of PET Patient level Classifications including estimates and CI of Sensitivity and Specificity according to each blinded reader. Frequencies will be displayed in a bar chart. Sensitivity and Specificity will be plotted for each reader including CI and performance goals.

### 4.14.3 Secondary Efficacy Variables

All secondary efficacy variables will be analyzed descriptively, with the exception of item 7; Kappa statistic.

Patient pathway through the study (PET scan, M0/M1, subsequent RP-PLND (Yes/No) and additional steps will be summarized and listed.

The following items are presented per secondary efficacy variable.

4.14.3.1 Percentage of patients in whom rhPSMA-7.3 (<sup>18</sup>F) imaging detects at least one verified M1 metastasis, as determined by central BIE.

This analysis concerns patients in the EEP with rhPSMA-7.3 (<sup>18</sup>F) imaging and confirmation tested (biopsy or additional imaging).

The percentage of patients with at least one M1 metastasis will be provided for each blinded independent reader. M1 metastasis requires the reader to identify a positive lesion in one of the three following locations: lymph nodes outside the pelvis, soft tissue/parenchyma or the bones. Patients will be counted to have M1 metastasis for this variable if a BIE detects M1 on the rhPSMA-7.3 (<sup>18</sup>F) and M1 is confirmed (biopsy, additional imaging) at the same location.

Patients where M1 was not verified (e.g. because the local reader did not detect M1) will be included in this analysis, as long as the BIE reader has detected M1 – in this case, the patients' metastasis will be considered as not verified. An additional table will be made using the EEP to summarize for each blinded reader the number of patients who have M1 by BIE and the presence / absence of confirmation of M1 metastasis.

TP-GDO-WW-016-07.a CONFIDENTIAL **Project Document Version No.** 3.0 Effective Date: 30 Jan 19 **Project Document Effective Date**: Date of last signature Related to: SOP-GDO-WW-019 

Blue Earth Diagnostics BED-PSMA-301

Statistical Analysis Plan

The endpoint for the secondary objective 1 of Verified Detection Rate (VDR) for M1 disease on a patient level is the percentage of patients with True-Positive M1 disease in the EEP.

VDR = (TP)/(TP+FP+TN+FN) where:

- TP = BIE PET positive and SoT positive
- FP = either: (1) BIE PET positive and SoT negative or (2) BIE PET positive and SoT not done or not proven (NB: If site PET = M0, we would still have baseline imaging and so will count in SoT)
- FN = BIE PET negative and SoT positive
- TN = either: (1) BIE PET negative and SoT negative or (2) BIE PET negative and SoT not done

Results for M1 detections by central, blinded readers will be reported overall and by SOT method used (histopathology, and imaging only) to confirm M1 detection as True Positive or False Positive.

4.14.3.2 Percentage of patients with negative conventional imaging for M1 disease in whom rhPSMA-7.3 (<sup>18</sup>F) PET detects at least one verified M1 metastasis, as determined by central BIE.

This analysis concerns patients in the EEP with rhPSMA-7.3 (<sup>18</sup>F) imaging and confirmation tested (biopsy or additional imaging) and with conventional imaging yielding negative M1 disease. The patients counted in this variable are a subset of 'Percentage of patients in whom rhPSMA-7.3 (<sup>18</sup>F) imaging detects at least one verified M1 metastasis, as determined by central BIE', where both the numerator and denominator are only counting patients with negative conventional imaging (according to investigator assessment) for M1 disease.

The endpoint for the secondary objective 2 of Verified Detection Rate (VDR) for M1 disease on a patient level with negative conventional imaging is the percentage of patients with negative conventional imaging (according to investigator assessment) for M1 disease and with True-Positive M1 disease according to rhPSMA-7.3 (<sup>18</sup>F) PET in the EEP.

4.14.3.3 Patient level PPV of rhPSMA-7.3 (<sup>18</sup>F) PET BIE for N1 and M1 lesions compared to histopathology or confirmatory imaging (M1 lesions only).

This analysis concerns EEP patients with rhPSMA-7.3 (<sup>18</sup>F) imaging and either N1 or M1 lesions detected.

PPV of N1 lesions is the proportion of patients with a positive PET BIE finding in pelvic lymph nodes and confirmed by histopathology, out of the patients with a positive PET BIE finding in pelvic lymph nodes.

PPV of M1 lesions is the proportion of patients with a positive PET BIE finding in other (extrapelvic) areas and confirmed by SoT (histopathology or confirmatory imaging (as determined by central SoT)), out of the patients with a positive PET BIE finding in other (extra-pelvic) areas.

TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019 CONFIDENTIAL Project Document Version No. 3.0

**Project Document Effective Date**: Date of last signature

Blue Earth Diagnostics BED-PSMA-301

Statistical Analysis Plan

4.14.3.4 PPV of rhPSMA-7.3 (<sup>18</sup>F) PET for detecting pelvic LN metastases compared to surgical pathology on a patient level in which a FP patient is defined as having at least one FP region (right or left pelvis), regardless of any coexisting TP findings.

This analysis concerns patients in the EAP where rhPSMA-7.3 (<sup>18</sup>F) imaging detected pelvic LN metastasis. Regions where rhPSMA-7.3 (<sup>18</sup>F) imaging detected no LN metastasis are not part of this by definition of PPV, hence only TP and FP regions will be taken into account.

$$PPV = TP / (TP + FP)$$

True positives will be all patients with a surgical pathology confirmed positive region and without a false positive region. False Positive patients will be those patients with any rhPSMA-7.3 (<sup>18</sup>F) PET positive region with negative surgical pathology or no surgical pathology.

4.14.3.5 NPV of rhPSMA-7.3 (<sup>18</sup>F) PET for detecting pelvic LN metastases compared to surgical pathology on a patient level in which a FN patient is defined as having at least one FN region (right or left pelvis), regardless of any coexisting TN findings.

This analysis concerns patients in the EAP with rhPSMA-7.3 (<sup>18</sup>F) imaging, where no LN metastases were detected and LN surgical pathology is available.

Regions where rhPSMA-7.3 (<sup>18</sup>F) imaging detected positive LN are not part of this by definition of NPV, hence only TN and FN regions will be taken into account.

$$NPV = TN / (TN + FN)$$

True negatives will be all patients with a surgical pathology confirmed negative region and without a false negative region. False negative patients will be those patients with any rhPSMA-7.3 (<sup>18</sup>F) PET negative region with positive surgical pathology.

### 4.14.3.6 Upstaging

- a) The percentage of patients being upstaged to N1 or M1 disease;
- b) The percentage of patients in whom planned RP is converted to EBRT.

The endpoints will be calculated as follows:

- Upstaging to N1 = Proportion of patients with positive BIE PET finding by BIE and negative conventional imaging finding from local investigator in pelvic lymph nodes, out of all the patients with evaluable scans.
- Upstaging to M1 = Proportion of patients with positive BIE PET finding and negative conventional imaging finding from local investigator in other (extra-pelvic) areas, out of all the patients with evaluable scans.

TP-GDO-WW-016-07.a CONFIDENTIAL Project Document Version No. 3.0 Effective Date: 30 Jan 19 Project Document Effective Date: Date of last signature Related to: SOP-GDO-WW-019 

Blue Earth Diagnostics BED-PSMA-301

Statistical Analysis Plan

- Planned RP converted to EBRT = Proportion of patients with positive BIE PET finding and planned RP changed to EBRT by local investigator, out of all the patients with evaluable scans.
- 4.14.3.7 Kappa statistic for the agreement between and within blinded independent readers on the interpretation of rhPSMA-7.3 (<sup>18</sup>F) scans.

This analysis concerns all EEP patients.

For this analysis, the patient's categorization to positive or negative by the blinded readers will be used, in pelvic lymph nodes and in extra-pelvic region.

## 4.14.3.7.1 Inter-reader agreement analysis

The Cohen's kappa statistic will be used to assess pairwise agreement between 2 readers including 95% exact CIs giving three kappa statistics (SAS® nomenclature: simple kappa). In addition, the Fleiss' kappa across the 3 readers including 95% (approximate) CIs will be shown (SAS® nomenclature: overall kappa Coefficient).

This same calculation will be repeated for the regions:

Prostate/Prostate Bed Pelvic Lymph Nodes Other

Other: Lymph nodes outside pelvis Other: Soft Tissue/parenchyma

Other: Bones.

### 4.14.3.7.2 Intra-reader agreement analysis

Cohen's Kappa will be used to assess intra-reader agreements in the first read and the repeat read of 10% of the randomly selected images for each of the three readers.

This same calculation will be repeated for the regions:

Prostate/Prostate Bed Pelvic Lymph Nodes Other

> Other: Lymph nodes outside pelvis Other: Soft Tissue/parenchyma

Other: Bones.

## 4.14.4 Exploratory Efficacy Variables

4.14.4.1 Diagnostic performance (sensitivity and specificity) of rhPSMA-7.3 (<sup>18</sup>F) PET for detecting pelvic LN metastases compared to surgical pathology on a regional level. This analysis will be performed using the EAP on all patients who were not diagnosed as M1 in the rhPSMA-7.3 (<sup>18</sup>F) PET imaging and for all sides where surgical pathology was performed.

TP-GDO-WW-016-07.a CONFIDENTIAL Project Document Version No. 3.0 Effective Date: 30 Jan 19 Project Document Effective Date: Date of last signature Related to: SOP-GDO-WW-019 

Blue Earth Diagnostics BED-PSMA-301

Statistical Analysis Plan

In this analysis, each patient will be considered as a cluster, with left hemi-pelvis and right hemi-pelvis considered as two observations within each cluster. Regions will be classified according to Table 3.

The descriptive parts of the primary analysis; cross table, sensitivity and specificity, will be repeated using region level analysis.

### 4.15 Safety Evaluation

All safety summaries and analyses will be based upon the FSP as defined in Section 4.5.

### 4.15.1 Adverse Events

For AEs and Serious AEs (SAEs), the MedDRA Version 22.1 or later will be used to code the reported events.

Treatment-emergent adverse events (TEAEs) will be tabulated and are defined as those AEs that either start or worsen in severity on or after the date/time of IP administration and on or before Day 4.

Where dates are missing or partially missing, AEs will be assumed to be treatment-emergent, unless there is clear evidence (through comparison of partial dates) to suggest that the AE started prior to IP administration or more than 4 days after IP administration.

In particular this means the following rules will be applied until a classification is given:

- 1. An AE with a missing start date and missing end date will be a TEAE
- 2. An AE with a missing start date and end date after IP administration will be TEAE
- 3. A start date with a missing year but month present will be assumed to have a year such that the start date is after informed consent and before Day 90. If these rules conflict then the rule 'after informed consent' prevails.
- 4. An AE will not be a TEAE if the start date is incomplete and
  - a. The end date of the AE is before the dosing date
  - b. The end date/time of an AE is before the dosing date/time
  - c. The day of the AE end date is missing and the month of the AE end date is before the month of dosing date
- 5. An AE will not be a TEAE if the AE start day of month is missing and
  - a. The last day of the AE start month is before the dosing date
  - b. The first day of the AE start month is more than 4 days after dosing

All AE summaries will provide the number of patients reporting at least one AE and the total number of events reported.

The following summaries will be provided:

• A summary of the number and percentage of patients reporting an AE, including counts of TEAEs, IP-related TEAEs, SAEs and IP-related SAEs.

TP-GDO-WW-016-07.a CONFIDENTIAL Project Document Version No. 3.0 Effective Date: 30 Jan 19 Project Document Effective Date: Date of last signature Related to: SOP-GDO-WW-019 

Blue Earth Diagnostics BED-PSMA-301

Statistical Analysis Plan

- A summary of the number and percentage of patients reporting a TEAE by SOC, and PT
- A summary of the number and percentage of patients reporting a TEAE by Common Terminology Criteria for Adverse Events (CTCAE) grade, SOC and PT
- A summary of the number and percentage of patients reporting a TEAE by causality, SOC and PT

Adverse event summaries will be ordered in terms of decreasing frequency for SOC, and PT within an SOC and then alphabetically for SOC, and PT within SOC.

For each patient and each adverse event, the worst CTCAE Toxicity grade (Version 5) recorded will be attributed and used in the by-severity summaries. Similarly, the worst causality (most related to treatment) will be attributed and used in the by-causality summaries. If CTCAE is missing for, the missing category will be used as worst category. If causality is missing, the worst case will be assumed.

A by-patient listing of all adverse events (including non-treatment-emergent events) will be provided. This listing will include center, patient identifier, age, race, adverse event (SOC, PT, and verbatim term), date of onset, date of resolution, duration, CTCAE, seriousness, action taken, outcome and causality.

### 4.15.2 Deaths, Serious Adverse Events, and Other Significant Adverse Events

Deaths, SAEs, and Other Significant AEs will be listed and summarized if numbers allow. The following summaries are planned.

- A summary of the number and percentage of TEAE leading to death
- A summary of the number and percentage of patients reporting a serious TEAE, by SOC and PT
- A summary of the number and percentage of patients with TEAEs leading to discontinuation of study treatment, by SOC and PT

The following listings will be created:

- A by-patient listing of all deaths that occurred during the study
- A by-patient listing of all SAEs
- A by-patient listing of all AEs leading to discontinuation of study treatment

Listings will follow the format described for AEs in Section 4.15.2.

### 4.15.3 Clinical Laboratory Evaluation

Blood safety laboratory values (hematology, biochemistry and coagulation) will be listed by patient and study time point including changes from baseline. The baseline for the laboratory values will be the pre-dose results obtained on Day 1.

TP-GDO-WW-016-07.a CONFIDENTIAL **Project Document Version No.** 3.0 Effective Date: 30 Jan 19 **Project Document Effective Date**: Date of last signature Related to: SOP-GDO-WW-019 

Blue Earth Diagnostics BED-PSMA-301

Statistical Analysis Plan

All values outside the clinical reference ranges will be flagged in the data listings. The abnormal values will be flagged with 'L' for values below the lower limit of the clinical reference range and 'H' for values above the upper limit of the clinical reference range and included in the listings.

Descriptive statistics (for non-categorical data including hematology and blood chemistry) will be presented for both individual values (N, mean, SD, median, minimum, maximum) and changes from baseline.

The following summaries will be provided:

- A summary of each laboratory parameter at visit 2 (pre-dose at day 1) and visit 3
- A summary of the change from baseline to visit 3 in each laboratory parameter
- A shift table of the number and percentage of patients experiencing treatment-emergent laboratory abnormalities at baseline vs visit 3, by laboratory parameter

### 4.15.4 Vital Signs, Physical Findings and Other Observations Related to Safety

Vital signs will be listed, including change from baseline. Baseline will be the last assessment before dosing, this is planned to be Visit 2 (Day 1), but may be any other assessment. A summary of each vital sign parameter, including change from baseline to visit 3 will be given.

12-lead ECG results will be listed, including change from baseline by patient and time point. Baseline will be the pre-dose assessment at Visit 2 (Day 1). A summary of each ECG parameter, including change from baseline to visit 3 will be given.

Physical examinations results (Normal, Abnormal Not Clinically Significant, Abnormal Clinically Significant) will be listed by patient and time point. Physical examination findings will be summarized by visit.

Heart rate category (<40 bpm, 40-59 bpm, 60-100 bpm, 101-130 bpm, >130 bpm) will be summarized and a shift table will be presented. Shift tables will be presented for OTc and physical examinations.

### 4.15.5 Other safety

A summary of injection site reactions during or immediately after the dose will be provided.

## 4.15.6 Safety Monitoring (Independent Data Monitoring Committee [IDMC], Data Monitoring Committee [DMC], Data and Safety Monitoring Board [DSMB])

Not applicable.

TP-GDO-WW-016-07.a CONFIDENTIAL Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019

**Project Document Version No. 3.0** 

**Project Document Effective Date**: Date of last signature


Blue Earth Diagnostics BED-PSMA-301

Statistical Analysis Plan

### 4.16 Determination of Sample Size

A total sample size of approximately 375 patients is planned in order to obtain 300 evaluable patients for analysis of the primary endpoint. Assuming a sensitivity of 40% of PSMA ligands for detecting N1 disease (based on the previous OSPREY [NCT02981368]), a sample size of 75 positive cases provides 90% power to reject the performance goal of 22.5%. Assuming a specificity of 90% for rhPSMA-7.3 (<sup>18</sup>F) PET, a sample size of 225 negative cases provides 90% power to reject the performance goal of 82.5%. Assuming the true prevalence rate of N1 disease is 25%, a sample size of 300 evaluable patients is expected to provide 75 positive cases and 225 negative cases.

Up to approximately 375 patients with unfavorable intermediate-, high- and very high-risk PCa will be enrolled into the study. Since some patients will have M1 disease and some patients will receive EBRT instead of RP following the PET scan, enrollment of up to approximately 375 patients will ensure inclusion of at least 300 evaluable patients undergoing RP and PLND.

In order to have sufficient numbers of histologically positive and negative cases, an interim look will be allowed to ensure a distribution of pN1 disease as would be anticipated in this patient population. After the inclusion of approximately 150 patients, the percentages of pN0 and pN1 will be monitored. If the percentage of pN1 exceeds 35%, inclusion of very high-risk and/or high-risk patients will be suspended. If the percentage of pN1 is less than 15%, the inclusion of intermediate-risk patients will be suspended.

## 4.17 Changes in the Conduct of the Study or Planned Analysis

An additional analysis set (Extended Efficacy Population) was created to accommodate analysis of patients where no RP and PLND was performed, such as patients with M1 lesions.

The second exploratory Efficacy objective and endpoint were removed. Objective:

To evaluate diagnostic performance of rhPSMA-7.3 ( $^{18}$ F) PET (as determined by central BIE) in patients with a) pelvic LN metastatic deposits <5 mm (short axis) and LN metastatic deposits  $\geq$ 5 mm (short axis) and b) pelvic LN metastatic deposits  $\leq$ 10 mm (short axis) and LN metastatic deposits  $\geq$ 10 mm (short axis), if feasible.

### Endpoint:

Diagnostic performance of rhPSMA-7.3 ( $^{18}$ F) PET in patients with a) pelvic LN metastatic deposits <5 mm (short axis) and LN metastatic deposits  $\geq$ 5 mm (short axis) and b) pelvic LN metastatic deposits  $\leq$ 10 mm (short axis) and LN metastatic deposits  $\geq$ 10 mm (short axis)

Two changes were documented to make the analysis description consistent.

• In Table 4 part b, which originated as table 6b in the CSP, the following text was changed: CSP: "Secondary analysis: PET is negative on True Positive (TP) region and PET is positive on True Negative (TN) region"

TP-GDO-WW-016-07.a CONFIDENTIAL Project Document Version No. 3.0 Effective Date: 30 Jan 19 Project Document Effective Date: Date of last signature Related to: SOP-GDO-WW-019 

Blue Earth Diagnostics BED-PSMA-301

Statistical Analysis Plan

SAP: "Secondary analysis: PET is negative in a histopathology positive region, and PET is positive in a histopathology negative region".

• In section 16.4 the text was adapted:

CSP: "Two analyses will be performed based on the classification of patients with one TP region and one TN region. The primary analysis will include patients as FN if they only had one positive region by histopathology and it was missed by PET. Full diagnostic statistics will be provided for both patient level classifications."

SAP will interpret this as: "Two analyses will be performed based on the classification of patients with one positive region and one negative region by histopathology. The primary analysis will include patients as FN if they only had one positive region by histopathology and it was missed by PET. Full diagnostic statistics will be provided for both patient level classifications."

### 5 REFERENCES

- [1] SAS® Version 9.3 of the SAS® System for Personal Computers. Copyright © 2011. SAS® Institute Inc. SAS® and all other SAS® Institute Inc. product or service names are registered trademarks or trademarks of SAS® Institute Inc., Cary, NC, USA.
- [2] Guidance for Industry and FDA Staff Statistical Guidance on Reporting Results from Studies Evaluating Diagnostic Tests. Available at: <a href="https://www.fda.gov/media/71147/download">https://www.fda.gov/media/71147/download</a> [Accessed 09 March 2020]
- [3] Jemal A, Bray F, Center MM, et al. Global cancer statistics. CA Cancer J Clin 2011;61(2):69-90
- [4] Klevečka V, Musch M, Roggenbuck U, et al. The incidence of lymph node metastases in prostate carcinoma depends not only on tumor characteristics but also on surgical performance and extent of pelvic lymphadenectomy. Medicina (Kaunas) 2008;44(8):601-8.
- [5] MSKCC, Nomogram. Available at: https://www.evidencio.com/models/show/440 [Accessed 23 January 2020].
- [6] NCCN Clinical Practice Guidelines in Oncology Prostate Cancer, 1.2020 16 March 2020.
- [7] OSPREY: Rowe S, Gorin M, Pienta K, et al. Results from the OSPREY trial: a prospective phase 2/3 multi-center study of <sup>18</sup>F-DCFPyL PET/CT imaging in patients with prostate cancer examination of diagnostic accuracy. J Nucl Med 2019;60(Suppl 1):586.

TP-GDO-WW-016-07.a CONFIDENTIAL **Project Document Version No.** 3.0 Effective Date: 30 Jan 19 **Project Document Effective Date**: Date of last signature Related to: SOP-GDO-WW-019 

Blue Earth Diagnostics BED-PSMA-301

Statistical Analysis Plan

- [8] Schulz KF, Altman DG, Moher D. CONSORT 2010 Statement: updated guidelines for reporting parallel group randomised trials. BMJ 2010;340:c332
- [9] UICC, TNM Classification of Malignant Tumors. Available at: https://www.uicc.org/resources/tnm [Accessed 23 January 2020]
- [10] Zhou XH, Obuchowski NA and McClish, DK. Statistical Methods in Diagnostic Medicine. Wiley, New York, 2002 pp 104-6

### 6 Appendix

### 6.1 SAS program to reproduce data in Zhou et al [10].

```
data one;
input TN
              No Polyps;
Cards;
       1
2
       2
1
       1
2
       2
2
       2
1
       1
1
       1
1
1
       1
2
       2
0
       1
2
       3
2
       2
1
       1
1
1
2
       2
       2
1
0
       2
1
       1
2
       2
2
2
       2
0
       1
;;;;
run;
proc sql;
   create table two as
      select
         No Polyps,
         TN/No Polyps as Sei hat,
          Se hat,
         No Polyps/mNo as Ni N,
          (calculated Ni N) * (calculated Ni N)
              * (calculated Sei hat-Se hat) * (calculated Sei hat-Se hat) as fc,
          sum(calculated fc) as sfc,
          calculated sfc/(n*(n-1)) as varSe hat
```

TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019 CONFIDENTIAL Project Document Version No. 3.0

Project Document Effective Date: Date of last signature


### Blue Earth Diagnostics

BED-PSMA-301 Statistical Analysis Plan

```
from
         (select
            sum(TN) as sTN,
            sum(No Polyps) as sNo,
            mean(No_Polyps) as mNo,
            count(*) as n,
            calculated sTN/calculated SNo as Se hat
            from one ) as o,
         one;
quit;
data final;
  set two;
  if n = 1;
  CI L = Se hat - (quantile('NORMAL', .975)*varSe hat**0.5);
  CI_U = Se_hat + (quantile('NORMAL', .975)*varSe_hat**0.5);
  p value = 1 - CDF('NORMAL', (Se hat-0.625)/varSe hat**0.5);
  keep Se_hat varSe_hat CI_L CI_U p_value;
run;
data final logit;
  set final;
   logit Se hat = log(Se hat/(1-Se hat));
   logit varSe hat = varSe hat*((1/(Se hat*(1-Se hat)))**2);
  logit_CI_L = logit_Se_hat - (quantile('NORMAL', .975)*logit_varSe_hat**0.5);
  logit_CI_U = logit_Se_hat + (quantile('NORMAL', .975)*logit_varSe_hat**0.5);
  logit zero one CI L = (CONSTANT('E') **logit CI L)/((CONSTANT('E') **logit CI L)+1);
  logit zero one CI U = (CONSTANT('E') **logit CI U)/((CONSTANT('E') **logit CI U)+1);
```

TP-GDO-WW-016-07.a Effective Date: 30 Jan 19 Related to: SOP-GDO-WW-019 CONFIDENTIAL Project Document Version No. 3.0

Project Document Effective Date: Date of last signature


## **DocuSign**

Status: Completed

**Timestamp** 

Sent: 01-Oct-2021 | 13:02

Viewed: 01-Oct-2021 | 13:26

Signed: 01-Oct-2021 | 13:27

Sent: 01-Oct-2021 | 13:02 Viewed: 01-Oct-2021 | 13:07

Signed: 01-Oct-2021 | 13:09

### **Certificate Of Completion**

Envelope Id: 06D06F4C86F7406B912081145A223308

Subject: Please DocuSign: BED\_PSMA\_301\_LIGHTHOUSE\_245596 SAP 3.0.pdf

Source Envelope:

Document Pages: 37 Signatures: 2 Envelope Originator:

Certificate Pages: 5 Initials: 0 Jane Silverwood

AutoNav: Enabled Via E. Folli, 50

AutoNav: Enabled Via E. Folli, 50
EnvelopeId Stamping: Enabled Milan, . 20134

Time Zone: (UTC+01:00) Amsterdam, Berlin, Bern, Rome, Stockholm, Vienna

Jane.Silverwood@blueearthdx.com

IP Address: 81.114.157.82

**Record Tracking** 

Status: Original Holder: Jane Silverwood Location: DocuSign

01-Oct-2021 | 13:00 Jane.Silverwood@blueearthdx.com

Signer Events
Albert Chau

albert.chau@blueearthdx.com Head of Biometrics (Interim)

Security Level: Email, Account Authentication

(Required)

Signature

Albert Chan

Signature Adoption: Pre-selected Style

Signature ID:

AF14745C-845B-4026-901B-623B25066E48

Using IP Address: 82.41.112.233

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I approve this document

**Electronic Record and Signature Disclosure:** 

Accepted: 07-Jun-2021 | 21:32 ID: 143372be-bf2f-42f4-81e1-eb97b2282108

Kees Duineveld

Kees.duineveld@parexel.com

Security Level: Email, Account Authentication

(Required)

— DocuSigned by:
Kees Duineveld

Signer Name: Kees Duineveld
Signing Reason: I am the author of this document
Signing Time: 01-Oct-2021 | 4:09:08 AM PDT
AC6BBDD8D7E04E2E9D735FC7C9119C6C

Signature Adoption: Pre-selected Style

Signature ID:

AC6BBDD8-D7E0-4E2E-9D73-5FC7C9119C6C

Using IP Address: 193.102.79.15

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I am the author of this document

**Electronic Record and Signature Disclosure:** 

Accepted: 01-Oct-2021 | 13:07

In Person Signer Events

ID: 83f7db16-0eb6-455d-ab5f-d354464bd1d4

Signature Timestamp

Editor Delivery Events Status Timestamp

Agent Delivery Events Status Timestamp

Intermediary Delivery Events Status Timestamp

| Certified Delivery Events | Status | Timestamp |
|---|---|---|
| Carbon Copy Events | Status | Timestamp |
| Witness Events | Signature | Timestamp |
| Notary Events | Signature | Timestamp |
| Envelope Summary Events | Status | Timestamps |
| Envelope Sent | Hashed/Encrypted | 01-Oct-2021 13:02 |
| Certified Delivered | Security Checked | 01-Oct-2021 13:07 |
| Certified Delivered Signing Complete | Security Checked Security Checked | 01-Oct-2021 13:07<br>01-Oct-2021 13:09 |
| | • | · |
| Signing Complete | Security Checked | 01-Oct-2021 13:09 |

### ELECTRONIC RECORD AND SIGNATURE DISCLOSURE

From time to time, Bracco Part 11 (we, us or Company) may be required by law to provide to you certain written notices or disclosures. Described below are the terms and conditions for providing to you such notices and disclosures electronically through the DocuSign system. Please read the information below carefully and thoroughly, and if you can access this information electronically to your satisfaction and agree to this Electronic Record and Signature Disclosure (ERSD), please confirm your agreement by selecting the check-box next to 'I agree to use electronic records and signatures' before clicking 'CONTINUE' within the DocuSign system.

### Getting paper copies

At any time, you may request from us a paper copy of any record provided or made available electronically to you by us. You will have the ability to download and print documents we send to you through the DocuSign system during and immediately after the signing session and, if you elect to create a DocuSign account, you may access the documents for a limited period of time (usually 30 days) after such documents are first sent to you. After such time, if you wish for us to send you paper copies of any such documents from our office to you, you will be charged a \$0.00 per-page fee. You may request delivery of such paper copies from us by following the procedure described below.

### Withdrawing your consent

If you decide to receive notices and disclosures from us electronically, you may at any time change your mind and tell us that thereafter you want to receive required notices and disclosures only in paper format. How you must inform us of your decision to receive future notices and disclosure in paper format and withdraw your consent to receive notices and disclosures electronically is described below.

## Consequences of changing your mind

If you elect to receive required notices and disclosures only in paper format, it will slow the speed at which we can complete certain steps in transactions with you and delivering services to you because we will need first to send the required notices or disclosures to you in paper format, and then wait until we receive back from you your acknowledgment of your receipt of such paper notices or disclosures. Further, you will no longer be able to use the DocuSign system to receive required notices and consents electronically from us or to sign electronically documents from us.

### All notices and disclosures will be sent to you electronically

Unless you tell us otherwise in accordance with the procedures described herein, we will provide electronically to you through the DocuSign system all required notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you during the course of our relationship with you. To reduce the chance of you inadvertently not receiving any notice or disclosure, we prefer to provide all of the required notices and disclosures to you by the same method and to the same address that you have given us. Thus, you can receive all the disclosures and notices electronically or in paper format through the paper mail delivery system. If you do not agree with this process, please let us know as described below. Please also see the paragraph immediately above that describes the consequences of your electing not to receive delivery of the notices and disclosures electronically from us.

### **How to contact Bracco Part 11:**

You may contact us to let us know of your changes as to how we may contact you electronically, to request paper copies of certain information from us, and to withdraw your prior consent to receive notices and disclosures electronically as follows:

To contact us by email send messages to: docusign.admin@bracco.com

### To advise Bracco Part 11 of your new email address

To let us know of a change in your email address where we should send notices and disclosures electronically to you, you must send an email message to us at docusign.admin@bracco.com and in the body of such request you must state: your previous email address, your new email address. We do not require any other information from you to change your email address.

If you created a DocuSign account, you may update it with your new email address through your account preferences.

### To request paper copies from Bracco Part 11

To request delivery from us of paper copies of the notices and disclosures previously provided by us to you electronically, you must send us an email to andrea.provini@bracco.com and in the body of such request you must state your email address, full name, mailing address, and telephone number. We will bill you for any fees at that time, if any.

### To withdraw your consent with Bracco Part 11

To inform us that you no longer wish to receive future notices and disclosures in electronic format you may:

i. decline to sign a document from within your signing session, and on the subsequent page, select the check-box indicating you wish to withdraw your consent, or you may;

ii. send us an email to docusign.admin@bracco.com and in the body of such request you must state your email, full name, mailing address, and telephone number. We do not need any other information from you to withdraw consent.. The consequences of your withdrawing consent for online documents will be that transactions may take a longer time to process..

### Required hardware and software

The minimum system requirements for using the DocuSign system may change over time. The current system requirements are found here: <a href="https://support.docusign.com/guides/signer-guide-signing-system-requirements">https://support.docusign.com/guides/signer-guide-signing-system-requirements</a>.

### Acknowledging your access and consent to receive and sign documents electronically

To confirm to us that you can access this information electronically, which will be similar to other electronic notices and disclosures that we will provide to you, please confirm that you have read this ERSD, and (i) that you are able to print on paper or electronically save this ERSD for your future reference and access; or (ii) that you are able to email this ERSD to an email address where you will be able to print on paper or save it for your future reference and access. Further, if you consent to receiving notices and disclosures exclusively in electronic format as described herein, then select the check-box next to 'I agree to use electronic records and signatures' before clicking 'CONTINUE' within the DocuSign system.

By selecting the check-box next to 'I agree to use electronic records and signatures', you confirm that:

- You can access and read this Electronic Record and Signature Disclosure; and
- You can print on paper this Electronic Record and Signature Disclosure, or save or send this Electronic Record and Disclosure to a location where you can print it, for future reference and access; and
- Until or unless you notify Bracco Part 11 as described above, you consent to receive exclusively through electronic means all notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you by Bracco Part 11 during the course of your relationship with Bracco Part 11.